CLINICAL TRIAL: NCT00816569
Title: Orthokeratology Contact Lenses for Keratoconus
Brief Title: Orthokeratology for Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: David Landau MD, : Hadassah Medical Organization, Jerusalem, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dvleyes-HMO-CTIL
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Orthokeratology; Keratoconus
Keywords: Orthokeratology; Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Keratoconus (Experimental): One eye of Keratoconus patient
  Interventions: Device: Orthokeratology contact lenses

INTERVENTIONS:
Device: Orthokeratology contact lenses — Wearing Orthokeratology lens in one eye of a keratoconus patient

SUMMARY:
To investigate a possible benefit of Orthokeratology contact lenses to improve uncorrected visual acuity of keratoconus patients

ELIGIBILITY:
Inclusion Criteria:

* Moderate Keratoconus
* No apical scars

Exclusion Criteria:

* Advanced Keratoconus
* Apical scaring
* Contact lens intolerance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual acuity | After 1 month

SECONDARY OUTCOMES:
Amount of change in corneal video-topography | At one month

CONTACTS AND LOCATIONS:
Locations (1):
- : Hadassah Medical Organization,, Jerusalem, Israel